CLINICAL TRIAL: NCT03495999
Title: Associations and Plausibility Among Left Ventricle Diastolic Function, Serum Uric Acid and Inflammatory Biomarkers in Individuals With Cardiometabolic Risks - A Prospective Observational Study
Brief Title: Hyperuricemia and Left Ventricular Diastolic Function
Status: Terminated | Type: Observational
Why Stopped: The study interest was reached
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Cheng-Wei Liu, Cardiologist, National Defense Medical Center, Taiwan
Other Study IDs: 2-106-05-078
Record Dates: First submitted 2018-04-03; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Hyperuricemia; Metabolic Syndrome; Left Ventricular Diastolic Dysfunction
Keywords: Hyperuricemia; Metabolic syndrome; Left ventricular diastolic dysfunction; Inflammation
MeSH Terms: conditions — Hyperuricemia; Metabolic Syndrome; Ventricular Dysfunction, Left; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normouricemia: Serum uric of 7mg/dl or less in men or 6mg/dl or less in women
  Interventions: Diagnostic Test: hyperuricemia
- Hyperuricemia: Serum uric of 7mg/dl or more in men or 6mg/dl or more in women
  Interventions: Diagnostic Test: hyperuricemia

INTERVENTIONS:
Diagnostic Test: hyperuricemia — serum uric acid of 7mg/dl or more in men or 6mg/dl or more in women

SUMMARY:
Metabolic syndrome and hyperuricemia were both associated with inflammation, leading to diversities of cardiovascular disease such as left ventricular diastolic dysfunction, but the relationship among these entities remained unclear. The aim of the present study focuses on the association among hyperuricemia, diastolic dysfunction and inflammatory biomarkers in apparently healthy individuals with metabolic syndrome

DETAILED DESCRIPTION:
Apparently healthy individuals with metabolic syndrome were prospectively and consecutively enrolled since August 2017. Blood samples were obtained after participants are fasting for at least 12 hours, including serum uric acid, high-sensitivity C-reactive protein, high-sensitivity interleukin-6, tumor necrotizing factor alpha, fasting glucose, glycosylated hemoglobin, insulin, lipid profile, creatinine, alanine aminotransferase, sodium, potassium, and calcium. All echocardiographic parameters were measured in accordance with the American Society of Echocardiography guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 75 years
2. Metabolic syndrome

Exclusion Criteria:

1. Left ventricular ejection fraction <40%
2. Severe valvular heart disease
3. Significant structure heart diseases such as hypertrophic, dilated, infiltrative or restrictive cardiomyopathy, or congenital heart disease
4. Persistent or chronic atrial fibrillation
5. Status post cardiac surgery, including coronary artery bypass surgery of valve intervention
6. Status post intra-cardiac device implantation
7. Chronic obstructive pulmonary disease
8. Severe anemia
9. An obvious systemic disease that interferes left ventricular diastolic dysfunction such as acute coronary syndrome

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Apparently healthy individuals with metabolic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Left ventricle diastolic dysfunction with elevated left atrial pressure | 1 day
  The contemporary definition of left ventricular diastolic dysfunction with elevated left atrial pressure is mainly >50% positive of the following criteria: (1) average E/e' ≥14 (2) left atrial volume index >34 ml/m2 (3) tricuspid regurgitation velocity >2.8 m/s

SECONDARY OUTCOMES:
high-sensitivity C-reactive protein | 1 week
  determined by Latex enhanced immunoturbidimetric，ADVIA 1800，ADVIA Chemistry XPT，Dimension RXL，SIEMENS，AU 640，Beckman Coulter
high-sensitivity interleukin-6 | 1 month
  determined by elisa enzyme-linked immunosorbent assay, R & D system
tumor necrotizing factor alpha | 1 month
  determined by elisa enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Wei Liu, M.D., Principal Investigator — Tri-service General hospital, Songshan branch, National defense medical center
Locations (1):
- Tri-service General Hospital, songshan branch, Taipei, Songshan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No